CLINICAL TRIAL: NCT06720038
Title: A Phase 2, Randomized, Double-Blind, Active-Controlled, Dose-Finding Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of VAX-31 in Healthy Infants Given 4 Doses at 2, 4, 6, and 12-15 Months of Age Concomitantly With Routine Pediatric Vaccines
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of VAX-31 in Healthy Infants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxcyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAX31-201
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Vaccines
Keywords: 31 Valent PCV; Pneumonia; Pneumococcal Infection
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- VAX-31 Low (Experimental): Participants will receive 4 doses of VAX-31 administered as an intramuscular injection at 2, 4, 6, and 12-15 months of age at one of four dose levels.
  Interventions: Biological: 0.5 mL of the low dose VAX-31
- VAX-31 Mid (Experimental): Participants will receive 4 doses of VAX-31 administered as an intramuscular injection at 2, 4, 6, and 12-15 months of age at one of four dose levels.
  Interventions: Biological: 0.5 mL of the mid dose VAX-31
- VAX-31 High (Experimental): Participants will receive 4 doses of VAX-31 administered as an intramuscular injection at 2, 4, 6, and 12-15 months of age at one of four dose levels.
  Interventions: Biological: 0.5 mL of the high dose VAX-31
- PCV20 (Active Comparator): Participants will receive 4 doses of PCV20 administered as an intramuscular injection of the standard dose at 2, 4, 6, and 12-15 months of age.
  Interventions: Biological: 0.5 mL dose of PCV20
- VAX-31 High-PFS (Experimental): Participants will receive 4 doses of VAX-31 administered as an intramuscular injection at 2, 4, 6, and 12-15 months of age at one of four dose levels.
  Interventions: Biological: 0.5 mL of the High-PFS dose VAX-31

INTERVENTIONS:
Biological: 0.5 mL of the low dose VAX-31 — 31 valent pneumococcal conjugate vaccine
  Arms: VAX-31 Low
Biological: 0.5 mL of the mid dose VAX-31 — 31 valent pneumococcal conjugate vaccine
  Arms: VAX-31 Mid
Biological: 0.5 mL of the high dose VAX-31 — 31 valent pneumococcal conjugate vaccine
  Arms: VAX-31 High
Biological: 0.5 mL dose of PCV20 — 20 valent pneumococcal conjugate vaccine
  Arms: PCV20
Biological: 0.5 mL of the High-PFS dose VAX-31 — 31 valent pneumococcal conjugate vaccine
  Arms: VAX-31 High-PFS

SUMMARY:
The objective of the study is to evaluate the safety, tolerability, and immunogenicity of 4 injections of VAX-31 (at 4 dose levels) compared to PCV20 in infants at 2, 4, 6, and 12-15 months of age, in addition to receiving routine US concomitant vaccines. Stage 1 of the study will comprise 3 dose ascending cohorts. Stage 2 of the study will enroll approximately 352 subjects. Stage 3 of the study will enroll approximately 500 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female infant ≥42 days to ≤89 days.
2. Full-term infant at least 37 weeks gestational age at birth.
3. Afebrile for ≥72 hours with an tympanic or rectal temperature <38.0°C (<100.4°F) before receipt of study vaccine.*Criterion applies to each vaccination. If not met, visit may be rescheduled for a time when no longer febrile for ≥72 hours.
4. Able to attend all scheduled visits and comply with the study procedures.
5. Subject's parent/legal guardian is able to read and understands the study procedures, alternate treatments, risks and benefits, and provides written informed consent.
6. Subject's parent/legal guardian is able to fill out an eDiary of solicited AE and take daily tympanic temperature and measurements of local injection site reactions for the 7 days after each study vaccination.
7. Subject's parent/legal guardian has an email address and access to a computer or smartphone with internet to complete the eDiary.

Exclusion Criteria:

1. History of invasive pneumococcal disease (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease.
2. Previous receipt of a licensed or investigational vaccine (excluding 1 dose of hepatitis B vaccine).
3. Known hypersensitivity to any vaccine.
4. Known or suspected impairment of immunological function (e.g., asplenia, human immunodeficiency virus, primary immunodeficiency).
5. Use of any immunosuppressive therapy or planned use through the last blood draw (Visit 6). Receipt of a <14-day course of systemic corticosteroids is not exclusionary if completed ≥1 month prior to first study vaccination. Topical and inhaled/nebulized steroids are also permitted.
6. History of failure to thrive or prior hospitalization for any chronic condition.
7. Subject has a bleeding disorder contraindicating IM vaccination.
8. Subject or his/her mother has documented hepatitis B surface antigen-positive test.
9. Subject has a known neurologic or cognitive behavioral disorder.
10. Subject has a known clinically significant congenital malformation or serious chronic disorder.
11. Receipt of a blood transfusion or blood products, including immunoglobulins.
12. Receipt of any investigational study product since birth, currently participating in another interventional investigational study, or plans to receive another investigational product while on study.
13. Any infant who cannot be adequately followed for safety according to the protocol plan.
14. Any other reason that in the opinion of the Investigator may interfere with the evaluation required by the study.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 905 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with any solicited local injection site adverse events (AE) within 7 days after each vaccination | 7 days after each vaccination
  Solicited local reactions include erythema, edema, and tenderness at the injection site
Percentage of subjects with any solicited systemic AE within 7 days after each vaccination | 7 days after each vaccination
  Solicited systemic reactions include fever, irritability, decreased appetite, decreased sleep, and increased sleep
Percentage of subjects with any unsolicited AE within 1 month after each vaccination | 1 months after each vaccination
  Percentage of subjects with unsolicited AE
Percentage of subjects with any medically attended adverse events (MAAE) within 6 months after last vaccination | 6 months after last vaccination
  Percentage of subjects with MAAE
Percentage of subjects with any Serious Adverse Events (SAE) within 6 months after last vaccination | 6 months after last vaccination
  Percentage of subjects with SAE
Percentage of subjects with any new onset of chronic illness (NOCI) within 6 months after last vaccination | 6 months after last vaccination
  Percentage of subjects with NOCI

SECONDARY OUTCOMES:
Percentage of subjects achieving a serotype-specific anti-pneumococcal IgG antibody concentration ≥0.35 mcg/mL 1 month after Dose 3 | 1 month after Dose 3
  Percentage of subjects achieving a serotype-specific anti-pneumococcal IgG antibody concentration ≥0.35 mcg/mL
Serotype-specific IgG antibody geometric mean concentration (GMC) 1 month after Dose 3 | 1 month after Dose 3
  Antibody geometric mean concentrations as measured by IgG for the 31 pneumococcal serotypes in VAX-31
Serotype-specific IgG antibody GMC 1 month after Dose 4 | 1 month after Dose 4
  Antibody geometric mean concentrations as measured by IgG for the 31 pneumococcal serotypes in VAX-31

CONTACTS AND LOCATIONS:
Locations (45):
- United States (42):
  - The Children's Clinic of Jonesboro, P.A, Jonesboro, Arkansas
  - Matrix Clinical Research, Gardena, California
  - Matrix Clinical Research, Los Angeles, California
  - Orange County Research Institute, Ontario, California
  - Center for Clinical Trials of San Gabriel, West Covina, California
  - Children's Hospital of Colorado - Dept. of Infectious Disease, Aurora, Colorado
  - SEC Clinical Research, Pensacola, Florida
  - PAS Research, Tampa, Florida
  - Clinical Research Prime, LLP, Idaho Falls, Idaho
  - Clinical Research Prime - Rexburg, Rexburg, Idaho
  - Kentucky Pediatrics/Adult Research, Bardstown, Kentucky
  - ACC Pediatric Research, Haughton, Louisiana
  - Complete Children's Health, Lincoln, Nebraska
  - Be Well Clinical Studies Nebraska, Lincoln, Nebraska
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Senders Pediatrics, South Euclid, Ohio
  - Cyn3rgy Research, Gresham, Oregon
  - UPMC Children's Community Pediatrics - Bass Wolfson, Cranberry, Cranberry Township, Pennsylvania
  - Allegheny Health & Wellness Pavilion West, Erie, Pennsylvania
  - UPMC Children's Community Pediatrics - Norwin, North Huntingdon, Pennsylvania
  - UPMC Children's Community Pediatrics South Hills-Jefferson Hills, Pittsburgh, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh - General Academic Pediatrics (GAP), Pittsburgh, Pennsylvania
  - UPMC Children's Community Pediatrics Bass Wolfson-Squirrel Hill, Pittsburgh, Pennsylvania
  - UPMC Children's Community Pediatrics-Castle Shannon, Pittsburgh, Pennsylvania
  - Tribe Clinical Research, LLC dba Neighbors Clinical Research, Charleston, South Carolina
  - Tribe Clinical Research/Parkside Pediatrics, Simpsonville, South Carolina
  - Proactive RGV LLC, Brownsville, Texas
  - Javara Inc. /Texas Health Care, PLLC, Dallas, Texas
  - Oak Cliff Research Company, Dallas, Texas
  - Kool Kids Pediatrics (Dynamed), Houston, Texas
  - Sunrise Pediatrics, Houston, Texas
  - Mercury Clinical Research - Pediatric Associates, Houston, Texas
  - University of Texas Medical Branch - Sealy Institute for Vaccine Sciences, Clinical Trials Program, League City, Texas
  - Pediatric Center/Neutra Life Sciences, Richmond, Texas
  - AMR - Layton, Layton, Utah
  - AMR - Cottonwood, Murray, Utah
  - AMR - Roy, Roy, Utah
  - AMR South Jordan, South Jordan, Utah
  - AMR - Syracuse, Syracuse, Utah
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC, Gordonsville, Virginia
  - Clinical Research Partners, LLC., Richmond, Virginia
- Puerto Rico (3):
  - Ponce Medical School Foundation Inc. / CAIMED Center, Ponce
  - BRCR Global Puerto Rico, San Juan
  - Caribbean Medical Research Center, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Vaxcyte is committed to providing access to anonymized data from the company's clinical trials for the purpose of legitimate scientific research. Requests for data may be addressed to datasharing@vaxcyte.com. Requests must be accompanied by a detailed analysis plan and will be reviewed for scientific validity. Data will be made available after initial product approval. Sharing of data may require execution of a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be shared after deidentification and made available starting 6 months after initial product approval.
Access Criteria: Criteria will depend on the specific proposal received and may include qualification of the scientific researchers, potential contribution to the research field, scientific rigor of statistical and analytical methods, and other criteria appropriate for the proposal.